CLINICAL TRIAL: NCT05845710
Title: Protection Against Emboli During caRotid Artery Stenting Using a Neuroguard IEP® Direct 3-in-1 Delivery System Comprised oF a pOst-dilation Balloon, integRated eMbolic Filter, and A Novel Carotid stEnt - the PERFORMANCE III Study
Brief Title: Direct Access Carotid Artery Stenting Using the Neuroguard IEP System (PERFORMANCE III)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Contego Medical, Inc. (Industry)
Collaborators: Yale Cardiovascular Research Group (Other); CardioMed Device Consultants, LLC (Industry); Advance Research Associates (Other); iMedNet (Unknown); AG Mednet (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CSP-1997
Record Dates: First submitted 2023-04-26; First posted 2023-05-06 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Carotid Stenosis; Carotid Artery Diseases
Keywords: carotid artery stent
MeSH Terms: conditions — Carotid Stenosis; Carotid Artery Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Neuroguard IEP Direct System (Experimental): The Neuroguard IEP® 3-in-1 Direct Carotid Stent and Post-Dilation Balloon System with Integrated Embolic Protection (Neuroguard IEP Direct System) is a combination self-expanding carotid artery stent, nitinol embolic protection filter, and post-dilation balloon. Neuroguard IEP Direct System is used with the Neuroguard Direct Access Kit which includes the Flow Redirection System.
  Interventions: Device: Neuroguard IEP Direct System

INTERVENTIONS:
Device: Neuroguard IEP Direct System — carotid artery stenting, direct access with blood flow redirection

SUMMARY:
The PERFORMANCE III study is a prospective, multicenter single-arm, open label study to evaluate the safety and effectiveness of the Neuroguard IEP® Direct System for the treatment of carotid artery stenosis in subjects at elevated risk for carotid endarterectomy (CEA).

Eligible patients greater than or equal to 20 years of age and less than or equal to 80 years of age, are those who have been diagnosed with either de-novo atherosclerotic or post CEA restenotic lesion(s) in the internal carotid arteries (ICA) or at the carotid bifurcation with greater than or equal to 50% stenosis if symptomatic or greater than or equal to 70% stenosis if asymptomatic.

DETAILED DESCRIPTION:
A prospective, multicenter single-arm, open label study to evaluate the safety and effectiveness of the Neuroguard IEP® Direct System for the treatment of carotid artery stenosis in subjects at elevated risk for adverse events following carotid endarterectomy (CEA). The Neuroguard IEP Direct System is a 3-in-1 carotid stent delivery system consisting of an angioplasty balloon, an integrated embolic protection device and a nitinol self-expanding stent loaded over the balloon and constrained by an outer sheath. Eligible patients greater than or equal to 20 years of age and less than or equal to 80 years of age, are those who have been diagnosed with either de-novo atherosclerotic or post CEA restenotic lesion(s) in the internal carotid arteries (ICA) or at the carotid bifurcation with greater than or equal to 50% stenosis if symptomatic or greater than or equal to 70% stenosis if asymptomatic.

Symptomatic subjects are defined as having stroke or transient ischemic attack (TIA) in the ipsilateral hemisphere supplied by the target vessel carotid lesion or ipsilateral transient monocular blindness (amaurosis fugax) within 180 days prior to the index procedure.

Subjects will be followed for 30 days post index procedure with additional follow up for subjects having a stroke or cranial nerve injury.

ELIGIBILITY:
General Inclusion Criteria

1. Male and non-pregnant, non-breastfeeding female subjects whose age is ≥ 20 or ≤ 82 years of age.
2. Subject is willing and capable of complying with and understands all study protocol requirements, including the specified follow-up visits, and can be contacted by telephone.
3. Subject has signed a written informed consent form that has been approved by the local governing Institutional Review Board (IRB) of the respective clinical site.
4. Subject is diagnosed with carotid artery stenosis treatable with carotid artery stenting via direct carotid access and is considered a high operative risk for carotid endarterectomy (CEA).
5. Subject is diagnosed with either:

   1. Symptomatic carotid stenosis ≥ 50% as determined by angiography, CTA, or duplex ultrasound. Symptomatic is defined as having stroke, transient ischemic attack (TIA) in the ipsilateral hemisphere supplied by the target vessel carotid lesion or ipsilateral transient monocular blindness (amaurosis fugax) within 180 days prior to the procedure; or
   2. Asymptomatic carotid stenosis ≥ 70% as determined by angiography, CTA, or duplex ultrasound.
6. Subject has a lesion located in the internal carotid artery (ICA) and/or common carotid artery (CCA).
7. Subject has a modified Rankin Scale of ≤ 2 at the time of procedure.
8. Females of child-bearing potential have a negative pregnancy test within 24 hours prior to the index procedure.
9. Subject is willing and able to take dual anti platelet therapy for a minimum of 30 days following the index procedure.
10. Subject meets at least one physiologic or one anatomic high-risk criteria.

Anatomic High-Risk Conditions for CEA

1. Target lesion at or above C2 (level of jaw). 2. Prior head and neck surgery in the region of the carotid artery. 3. Tracheostomy or tracheostoma. 4. Surgically inaccessible lesion or hostile neck which the investigator deems safe for direct carotid access including but not limited to:

1. Prior neck irradiation
2. Radial neck dissection
3. Cervical spine immobility 5. Prior ipsilateral CEA. 6. Prior cranial nerve injury. 7. Severe tandem lesions. 8. Occlusion of the contralateral CCA or ICA. 9. Severe bilateral ICA stenosis.

   Physiological High-Risk Conditions for CEA
   1. Subject is ≥ 70 years of age (maximum 80 years) at the time of enrollment.
   2. Subject has NYHA Class III or IV congestive heart failure (CHF).
   3. Subject has chronic obstructive pulmonary disease (COPD) with FEV1 < 50, on intermittent or chronic oxygen therapy, or a resting PO2 of ≤ 60 mmHg (room air).

   4 Subject has left ventricular ejection fraction (LVEF) ≤ 35%. 5. Subject has angina class 3 or 4 or unstable angina. 6. Subject has a history of recent myocardial infarction (between 30 days and 6 weeks prior to index the procedure).

   7. Subject has coronary artery disease with two or more vessels with ≥ 70% stenosis.

   8. Subject has planned coronary artery bypass grafting (CABG) or peripheral vascular surgery between 31 and 60 days after index procedure.

   9. Subject has restenosis following a prior carotid endarterectomy (CEA).

   Angiographic Inclusion Criteria
   1. Subject has a lesion located in the internal carotid artery (ICA) and/or common carotid artery (CCA).
   2. Single de novo or restenotic (post carotid endarterectomy [CEA]) target lesion or severe tandem lesions that can be covered by a single Neuroguard stent.
   3. Target lesion is treatable with a single stent of up to 40 mm in length.
   4. Index vessel diameter (segment covered by the mid-portion of the stent) is between 4.0 mm and 6.0 mm at the site of the target lesion.
   5. Distal vessel diameter at the site of Neuroguard filter deployment is between 4.0 mm and 7.0 mm.
   6. Distal common carotid artery diameter (segment covered by proximal portion of the stent) is between 4.0 mm and 8.0 mm.
   7. Sufficient landing zone exists in the cervical internal carotid artery distal to the target lesion to allow for the safe and successful deployment of the integrated Neuroguard filter.
   8. At least 5 cm of atherosclerosis free space in the ipsilateral common carotid artery between the sheath insertion site and the proximal edge of the target lesion.
   9. Common carotid artery reference diameter is at least 6 mm.
   10. Target vessel must meet diameter requirements as set forth in the Neuroguard IEP Direct System Instructions for Use (IFU).

   General Exclusion Criteria
   1. Life expectancy of less than one year in the opinion of the investigator at the time of enrollment.
   2. Currently requiring an organ transplantation.
   3. An evolving acute stroke
   4. Anticipated or existing potential sources of emboli including left ventricular aneurysm, aortic or mitral mechanical heart valve, severe calcific aortic stenosis (valve area < 1.0 cm2), endocarditis, moderate to severe mitral stenosis, known previously symptomatic patent foramen ovale (PFO), left atrial thrombus, any intracardiac mass.
   5. Deep being thrombosis (DVT) or pulmonary embolism (PE) treated within the past 12 months.
   6. Recently (< 60 days) implanted heart valve.
   7. Subject has experienced any episode of paroxysmal atrial fibrillation or atrial flutter within the past 6 months or has a history of paroxysmal atrial fibrillation or atrial flutter requiring chronic anticoagulation.
   8. History of chronic atrial flutter or chronic atrial fibrillation.
   9. Anticoagulation with Phenprocoumon (Marcumar®), warfarin, direct thrombin inhibitors, or anti-Xa agents within 14 days of the index procedure.
   10. Subject with a known hypercoaguable state.
   11. Acute febrile illness (temperature ≥ 100.4°F or 38°C) or active infection.
   12. Subject with a SARS-CoV-2/COVID-19 infection within 21 days prior to the index procedure.
   13. Acute myocardial infarction < 30 days prior to index procedure.
   14. Any major surgical procedure (i.e., intraabdominal or intrathoracic surgery or any surgery / interventional procedure involving cardiac or vascular system) 30 days prior to or within 30 days following the index procedure.
   15. History of disabling stroke with substantial residual disability (modified Rankin score ≥ 3).
   16. Subject has had a transient ischemic attack (TIA) or amaurosis fugax within 48 hours prior to the index procedure.
   17. Known severe carotid stenosis contralateral to the target lesion requiring treatment within 30 days of the index procedure.
   18. Any other neurological deficit not due to stroke that may confound neurological assessments.
   19. Subject has contralateral laryngeal or vagus nerve injury.
   20. Subject has severe dementia.
   21. Subject has intracranial tumor.
   22. Known hypersensitivity to nitinol or its components (e.g., nickel, titanium).
   23. History of intracranial hemorrhage within the 12 months prior to the index procedure.
   24. History of gastrointestinal (GI) bleed within 30 days prior to the index procedure that would interfere with antiplatelet therapy.
   25. Any condition that precludes proper angiographic assessment or makes direct carotid artery access unsafe (e.g., severe hepatic impairment, malignant hypertension, morbid obesity).
   26. Subject has less than 5 cm between the direct carotid access site and the proximal edge of the target lesion.
   27. Known hypersensitivity to contrast media that cannot be adequately premedicated.
   28. Hemoglobin (Hgb) < 8 gm/dL, platelet count < 100,000, international normalized ratio (INR) > 1.5 (irreversible), or heparin-induced thrombocytopenia.
   29. Chronic renal insufficiency (serum creatinine > 2.5 mg/dL or estimated GFR < 30 cc/min) or end-stage renal disease on hemodialysis on the day of the index procedure.
   30. History or current indication of bleeding diathesis or coagulopathy including thrombocytopenia or an inability to receive heparin in amounts sufficient to maintain an activated clotting time (ACT) at ≥ 250 seconds, or uncorrectable severe anemia.
   31. Contraindication, intollerance or allergy to standard of care study medications, including antiplatelet therapy or aspirin.
   32. Previously enrolled in this study or currently enrolled in another interventional device or drug study that has not yet reached the primary endpoint.
   33. Potential for subject non-compliance with protocol-required follow up or antiplatelet medication in the opinion of the investigator.
   34. Subject is otherwise unsuitable for intervention or surgery in the opinion of the investigator.

   Angiographic Exclusion Criteria
   1. Total occlusion of the target carotid artery.
   2. Previously placed stent in the target vessel or the planned arteriotomy site.
   3. Excessive circumferential calcification of the target lesion, defined as > 3 mm of thickness of calcification seen in orthogonal views on fluoroscopy or on CTA.
   4. Qualitative characteristics of ipsilateral common carotid artery, ipsilateral external carotid artery, or target lesion that preclude or make difficult the safe introduction of the direct access sheath.
   5. Angiographic evidence of a mobile filling defect or fresh thrombus in the target carotid artery.
   6. Presence of "string sign" of the target lesion (a sub-totally occluded, long segment of the true lumen of the artery with markedly reduced contrast flow).
   7. Non-atherosclerotic carotid stenosis (e.g., dissection, fibromuscular dysplasia).
   8. Proximal/ostial CCA stenosis ≥ 50% or intracranial stenosis more severe than the target lesion.
   9. Subject in whom direct carotid access is not possible, including severe tortuosity or stenosis that requires additional endovascular procedures or that prevents safe and expeditious vascular access.
   10. Subject with intracranial pathology, that in the opinion of the investigator, makes the patient inappropriate for study participation (e.g., arteriovenous malformation, intracranial tumor, microangiopathy or large vessel cerebral vascular disease, etc.) or that would confound the neurological evaluation.
   11. Angiographic, CT, MR or ultrasound evidence of atherosclerosis of the common carotid artery that would preclude or make difficult safe placement of the sheath and other endovascular devices to the target artery as needed for carotid stenting.
   12. Angiographic, CT, MR or ultrasound evidence of severe tortuosity of the cervical internal carotid artery. Severe vascular tortuosity is defined as 2 or more bends of 90 degrees or more within 4 cm of the target lesion.
   13. Angiographic, CT, MR or ultrasound evidence of angulation or tortuosity (≥ 90 degree) of the common carotid artery (CCA) that will transmit a severe loop to the internal carotid after sheath placement.
   14. Subject with > 50% stenosis in the common carotid artery (CCA) proximal to the target lesion.

Ages: 20 Years to 82 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 178 (Actual)
Dates: Start 2023-10-05 (Actual); Primary Completion 2025-08-12 (Actual); Study Completion 2025-08-12 (Actual)

PRIMARY OUTCOMES:
Composite of Major Adverse Events (MAE) | Within 30 days of the study procedure
  The primary endpoint is a composite 30-day rate of Major Adverse Events (MAE), defined as the cumulative incidence of all stroke, myocardial infarction (MI) and death within 30 days of the index procedure.

SECONDARY OUTCOMES:
Acute Success | Procedure
  The ability to insert the Neuroguard IEP Direct System, deliver the stent, and remove the stent delivery catheter.
Technical Success | Procedure
  The ability to utilize the accessories provided in the Neuroguard Direct Access Kit to establish flow reversal, defined as visualization of blood in the collection tubing.
Procedure Success | Procedure
  Acute Success and Technical Success in the absence of device related Major Adverse Events (defined as the cumulative incidence of all stroke, myocardial infarction and death) prior to discharge.
Blood Transfusion | Procedure through discharge or within 30 days of the study procedure
  Number of subjects requiring blood transfusion from procedure initiation through to discharge.
Stroke, Death | Within 30 days of the study procedure
  Ipsilateral, major and minor stroke, all death, cardiac death, neurological death

CONTACTS AND LOCATIONS:
Overall Officials: Sean Lyden, MD, Principal Investigator — The Cleveland Clinic; D. Christopher Metzger, MD, Principal Investigator — OhioHealth Research Institute
Locations (32):
- United States (30):
  - Honor Health, Scottsdale, Arizona
  - Hartford Hospital, Hartford, Connecticut
  - MedStar Washington Hospital Center, Washington D.C., District of Columbia
  - Manatee Memorial Hospital, Bradenton, Florida
  - Delray Medical Center, Delray Beach, Florida
  - Mount Sinai Vascular Institute, Miami Beach, Florida
  - AdventHealth Orlando, Orlando, Florida
  - Indiana University Methodist Hospital, Indianapolis, Indiana
  - Southcoast Health, New Bedford, Massachusetts
  - McLaren Center for Research and Innovation, Bay City, Michigan
  - Hackensack University Medical Center, Hackensack, New Jersey
  - University at Buffalo Neurosurgery - Jacobs Institute, Buffalo, New York
  - Sisters of Charity Hospital, Buffalo, New York
  - Northwell Health, Lake Success, New York
  - Mount Sinai Medical Center, New York, New York
  - UNC Hospital, Chapel Hill, North Carolina
  - Atrium Health - Sanger Heart and Vascular, Charlotte, North Carolina
  - North Carolina Heart and Vascular Research, Raleigh, North Carolina
  - TriHealth (Bethesda North Hospital), Cincinnati, Ohio
  - Cleveland Clinic, Cleveland, Ohio
  - OhioHealth Research Institute, Columbus, Ohio
  - St. Francis Hospital, Tulsa, Oklahoma
  - Allegheny General Hospital, Pittsburgh, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Prisma Health, Greenville, South Carolina
  - Vanderbilt University, Nashville, Tennessee
  - St. David's Healthcare, Austin, Texas
  - Baylor Scott and White Research Institute, Dallas, Texas
  - UT Southwestern Medical Center, Dallas, Texas
  - Sentara Norfolk General Hospital, Norfolk, Virginia
- France (2):
  - Hopital Marie Lannelongue, Le Plessis-Robinson
  - GH Paris St. Joseph, Paris